CLINICAL TRIAL: NCT02240576
Title: Possible Manifestation of Rhinitis After Nasal Fracture
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57183
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Nasal Fracture
Keywords: surgery for nasal fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We would like to investigate our hypothesis of a higher prevalence of nasal fracture in the history of idiopathic rhinitis (IR) patients compared to healthy controls. Therefore a retrospective analysis of 310 patients with a nasal fracture in the past would be useful to investigate the incidence of IR in this cohort afterwards (5-10 y later).

DETAILED DESCRIPTION:
The patient population will be recruited by sending patient questionnaires (form in addendum) to patients who suffered a nasal fracture five to ten years ago (time period 2005-2013) with nose reposition afterwards under general anaesthesia in the chirurgical day care centre (CDC) of university hospital (UZ) Leuven.

The control population (HC) will be recruited by sending a slightly adapted questionnaire (form in addendum) to patients who had surgery of the vocal cords under general anaesthesia in the CDC of UZ Leuven in the same period as the patient group. The control group will be age and sex-matched with the patient group.

ELIGIBILITY:
Inclusion Criteria:

* Presence of nasal fracture in 2005-2013 and
* Diagnosis ascertained by a Ear-Nose-Throat (ENT) specialist and
* Followed by nose reposition surgery under general anaesthesia and
* Described in the clinical operation report as "mobile nose bones" OR Available radiography

Inclusion criteria of the control group:

* Presence of problem on vocal cords without previous nasal fracture
* Surgery of the vocal cords under general anaesthesia in 2005-2013

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who suffered a nasal fracture five to ten years ago (time period 2005-2013) with nose reposition afterwards under general anaesthesia in the chirurgical day care centre (CDC) of Gasthuisberg.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the incidence of IR after nasal fracture in the patient population with the incidence of IR in the control group. | at least 1 year after surgery
  Comparison of the incidence of IR after nasal fracture in the patient population with the incidence of IR in the control group.
  outcome measurement: percentage of participants

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, Prof Dr, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven ENT, Leuven, Vlaams Brabant, Belgium